CLINICAL TRIAL: NCT07078773
Title: Application of Pericapsular Nerve Group (PENG) Block in Transurethral Resection of Bladder Tumors
Brief Title: Application of Pericapsular Nerve Group (PENG) Block
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Shi, associate professor, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20240724-01
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: TURBT
Keywords: Pericapsular Nerve Group (PENG) block; obturator nerve reflex
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG Group:Ultrasound-guided pericapsular nerve group (PENG) block. (Experimental): A convex ultrasound probe (frequency 2-5 MHz) was positioned at the patient's inguinal ligament, with one end directed toward the anterior inferior iliac spine (AIIS), clearly visualizing the bony prominences of the iliopubic eminence and the AIIS. The needle tip was directed medially toward the pectineus muscle. Upon reaching the space between the pectineus muscle and the pubic bone, and after confirming the absence of blood on aspiration, 30 ml of 0.375% ropivacaine was injected.
  Interventions: Procedure: peng block
- Control group : Ultrasound-guided obturator nerve block. (Active Comparator): An ultrasound probe was positioned at the inguinal ligament, with the needle inserted parallel to the long axis of the probe. After confirming no blood upon aspiration, 15 ml of 0.375% ropivacaine was injected into the fascial plane between the adductor brevis and adductor magnus, as well as into the midportion of the adductor longus and adductor brevis muscles.
  Interventions: Procedure: obturator nerve block

INTERVENTIONS:
Procedure: peng block — A convex ultrasound probe (frequency 2-5 MHz) was positioned at the patient's inguinal ligament, with one end directed toward the anterior inferior iliac spine (AIIS), clearly visualizing the bony prominences of the iliopubic eminence and the AIIS. The needle tip was directed medially toward the pectineus muscle. Upon reaching the space between the pectineus muscle and the pubic bone, and after confirming the absence of blood on aspiration, 30 ml of 0.375% ropivacaine was injected.
  Arms: PENG Group:Ultrasound-guided pericapsular nerve group (PENG) block.
Procedure: obturator nerve block — An ultrasound probe was positioned at the inguinal ligament, with the needle inserted parallel to the long axis of the probe. After confirming no blood upon aspiration, 15 ml of 0.375% ropivacaine was injected into the fascial plane between the adductor brevis and adductor magnus, as well as into the midportion of the adductor longus and adductor brevis muscles.
  Arms: Control group : Ultrasound-guided obturator nerve block.

SUMMARY:
This study aims to determine the efficacy and safety of the Pericapsular Nerve Group (PENG) block in preventing obturator nerve reflex during transurethral resection of bladder tumors.

DETAILED DESCRIPTION:
During transurethral resection of bladder tumors (TURBT), obturator nerve reflex is easily triggered during electrocautery. Currently, two primary methods are used to prevent obturator nerve reflex: deep neuromuscular blockade under general anesthesia and obturator nerve block. To date, no studies have confirmed the efficacy of the Pericapsular Nerve Group (PENG) block in preventing obturator nerve reflex.

This study recorded the percentage decrease in adductor muscle strength at various time points after the PENG block, the occurrence of intraoperative adductor muscle spasms, the duration of nerve block procedure, and the incidence of postoperative adverse events. The completion of this study could provide clinical evidence for selecting anesthesia methods in TURBT procedures and offer robust evidence-based support for relevant medical decisions by government health agencies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Scheduled for TURBT for unilateral bladder tumor;
* Able to understand and provide informed consent;

Exclusion criteria:

* Patients who refuse or are unable to provide informed consent;
* Allergic to local anesthetics, insensitive to propofol or general anesthetics;
* Pregnant women;
* Severe liver dysfunction;
* Evidence of infection at or near the proposed puncture site;
* Any sensory or motor impairment of the lower limbs;
* Recent (within 6 months) lower limb joint replacement surgery.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-07-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the percentage reduction in adductor muscle strength at 5, 10, 15, 20, 25, 30 minutes, and 3 hours after drug administration, compared to pre-administration levels. | 5, 10, 15, 20, 25, 30 minutes, and 3 hours post-administration
  The percentage increase in adductor strength from preoperative to postoperative measurements divided by preoperative adductor strength is larger, reflecting a better nerve block effect and superior obturator nerve reflex inhibition.

SECONDARY OUTCOMES:
Presence of obturator nerve reflex during surgery | During surgery
  Obturator nerve reflex grading system: No response in the adductor muscle group of the thigh; mild muscle twitching in the adductor muscle group of the thigh; severe contraction of the adductor muscle group of the thigh

OTHER OUTCOMES:
Physician Satisfaction Score | Up to 48 hours postoperative
  Grading:
  Excellent (1 point) Good (2 points) Fair (3 points) Poor (4 points) Higher scores indicate superior inhibition of obturator nerve reflex and better block efficacy
Incidence of adverse reactions such as local anesthetic toxicity and nerve injury post-administration. | Up to 48 hours postoperative
  The lower the incidence of adverse reactions such as local anesthetic toxicity and nerve injury, the better the PENG block technique. quantifies safety profile (lower incidence indicates higher safety)
Surgical Duration | During surgery
  Indirectly reflects interference from obturator nerve reflex; shorter duration implies effective reflex suppression
Needle Pass Count | During nerve block procedures
  Fewer passes indicate simpler operation and higher precision.
Operational Duration of Nerve Block | During nerve block procedures
  Reflects procedural convenience; shorter duration indicates simpler technique
Patient Satisfaction Score Patient Satisfaction Score Patient Satisfaction Score | Up to 48 hours postoperative
  Grading:
  Excellent (1 point) Good (2 points) Fair (3 points) Poor (4 points) Higher scores reflect enhanced patient comfort during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Liu Han, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshida T, Nakamoto T, Kamibayashi T. Ultrasound-Guided Obturator Nerve Block: A Focused Review on Anatomy and Updated Techniques. Biomed Res Int. 2017;2017:7023750. doi: 10.1155/2017/7023750. Epub 2017 Feb 9. PMID 28280738
- [Background] Bolat D, Aydogdu O, Tekgul ZT, Polat S, Yonguc T, Bozkurt IH, Sen V, Okur O. Impact of nerve stimulator-guided obturator nerve block on the short-term outcomes and complications of transurethral resection of bladder tumour: A prospective randomized controlled study. Can Urol Assoc J. 2015 Nov-Dec;9(11-12):E780-4. doi: 10.5489/cuaj.3149. Epub 2015 Nov 4. PMID 26600884
- [Background] Anagnostopoulou S, Kostopanagiotou G, Paraskeuopoulos T, Chantzi C, Lolis E, Saranteas T. Anatomic variations of the obturator nerve in the inguinal region: implications in conventional and ultrasound regional anesthesia techniques. Reg Anesth Pain Med. 2009 Jan-Feb;34(1):33-9. doi: 10.1097/AAP.0b013e3181933b51. PMID 19258986
- [Background] Turner K, Levi Sandri GB, Boucher E, Henno S, Le Prise E, Meunier B, Boudjema K, Sulpice L. Complete radiological response of an initially locally advanced unresectable pancreatic cancer to chemoradiotherapy using FOLFIRINOX regimen: report of a case. Clin Res Hepatol Gastroenterol. 2015 Apr;39(2):e29-31. doi: 10.1016/j.clinre.2014.08.011. Epub 2014 Oct 3. No abstract available. PMID 25288453
- [Background] Nielsen TD, Moriggl B, Soballe K, Kolsen-Petersen JA, Borglum J, Bendtsen TF. A Cadaveric Study of Ultrasound-Guided Subpectineal Injectate Spread Around the Obturator Nerve and Its Hip Articular Branches. Reg Anesth Pain Med. 2017 May/Jun;42(3):357-361. doi: 10.1097/AAP.0000000000000587. PMID 28263244

DOCUMENTS (1):
  • Study Protocol (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT07078773/Prot_000.pdf